CLINICAL TRIAL: NCT05657522
Title: Short-term Soft and Hard Tissue Changes Following Skeletal Anterior Open Bite Treatment Using the Rapid Molar Intruder
Brief Title: Early Treatment of Anterior Open Bite Using the Rapid Molar Intruder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-Ortho-17-2022
Record Dates: First submitted 2022-12-11; First posted 2022-12-20 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Open Bite
Keywords: Anterior open bite; Rapid molar intruder; Mixed dentition
MeSH Terms: conditions — Open Bite

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rapid Molar Intruder (Experimental): Patients in this group will undergo the interventional procedure, which is the application of the rapid molar intruder appliance. This will help in correcting the open bite.
  Interventions: Device: Rapid molar intruder
- Untreated Control Group (No Intervention): Patients in this group will be monitored without any active treatment.

INTERVENTIONS:
Device: Rapid molar intruder — The rapid molar intruder was applied.
  Arms: Rapid Molar Intruder

SUMMARY:
This study evaluated the efficacy of rapid molar intruder (RMI) in treating anterior open bite in the mixed dentition. The study sample consisted of 40 patients who had a skeletal anterior open bite. The sample was allocated randomly into two groups: the RMI group and the control group. The skeletal, dentoalveolar and soft tissue changes occurring after treatment were assessed by using lateral cephalometric images.

DETAILED DESCRIPTION:
Many appliances have been used to treat skeletal anterior open bite (AOB) malocclusion, such as removable appliances, extra-oral appliances (vertical chin cup and vertical head gear), fixed appliances, Orthognathic surgery and functional appliances. Treatment with these appliances produces soft and hard dentofacial tissue changes. Many studies have been carried out in order to study these changes.

In this study, the investigators treated AOB using RMI. Patients were divided into two groups to evaluate the efficacy of RMI.

RMI group: Rapid molar intruder was applied. Control group: Untreated control group. In order to evaluate the changes occurring, lateral cephalometric images were taken in both groups at the beginning of the treatment (T1) and after 9 months of the first cephalograms (T2).

ELIGIBILITY:
Inclusion Criteria:

1. Patients in the mixed dentition
2. Chronological age between 8 and 12 years
3. skeletal class I or II malocclusion
4. Skeletal anterior open bite was assessed clinically and then confirmed radiographically: SN/GoMe was greater than 33°, MM was greater than 27
5. No general problems
6. Good oral health

Exclusion Criteria:

1. Presence of periodontal diseases
2. Presence of general diseases, syndromes or cleft lip and palate
3. Patients with previous orthodontic treatment

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2013-09-25 (Actual); Primary Completion 2014-04-20 (Actual); Study Completion 2015-01-20 (Actual)

PRIMARY OUTCOMES:
Change in the SNA angle | Time 1: One week before the beginning of the treatment, Time 2: after nine months from the beginning of active treatment.
  Lateral cephalometric images were taken for each patient, and this angle was measured in degrees. This angle represents the position of the upper jaw in the cephalometric analysis in the anteroposterior direction.
Change in the SNB angle. | Time 1: One week before the beginning of the treatment, Time 2: after nine months from the beginning of active treatment.
  Lateral cephalometric images were taken for each patient, and this angle was measured in degrees. This angle represents the position of the lower jaw in the cephalometric analysis in the anteroposterior direction.
Change in the ANB angle | Time 1: One week before the beginning of the treatment, Time 2: after nine months from the beginning of active treatment.
  Lateral cephalometric images were taken for each patient, and this angle was measured in degrees. This angle represents the spatial relationship between the upper and lower jaws in the cephalometric analysis in the anteroposterior direction.
Change in the MM angle | Time 1: One week before the beginning of the treatment, Time 2: after nine months from the beginning of active treatment.
  Lateral cephalometric images were taken for each patient, and this angle was measured in degrees. This angle represents the amount of vertical divergence between the upper and lower jaws in the cephalometric analysis.
Change in the SN-OCP angle | Time 1: One week before the beginning of the treatment, Time 2: after nine months from the beginning of active treatment.
  Lateral cephalometric images were taken for each patient, and this angle was measured in degrees. This angle represents the relationship between the occlusion plane and the cranial base in the cephalometric analysis in the vertical direction.
Change in the SN-MP angle | Time 1: One week before the beginning of the treatment, Time 2: after nine months from the beginning of active treatment.
  Lateral cephalometric images were taken for each patient, and this angle was measured in degrees. This angle represents the relationship between the lower jaw plane and the cranial base in the cephalometric analysis in the vertical direction.
Change in the SN-SPP angle | Time 1: One week before the beginning of the treatment, Time 2: after nine months from the beginning of active treatment.
  Lateral cephalometric images were taken for each patient, and this angle was measured in degrees. This angle represents the relationship between the upper jaw plane and the cranial base in the cephalometric analysis in the vertical direction.
Change in the overbite (Ovb) | Time 1: One week before the beginning of the treatment, Time 2: after nine months from the beginning of active treatment.
  Lateral cephalometric images were taken for each patient. This was measured in millimetres vertically from the upper to the lower central incisors.
Change in the overjet (Ovj) | Time 1: One week before the beginning of the treatment, Time 2: after nine months from the beginning of active treatment.
  Lateral cephalometric images were taken for each patient. This was measured in millimetres Horizontally from the upper to the lower central incisors.
Change in the Bjork sum (NS-Ar + S-Ar-Go +Ar-Go-Me) | Time 1: One week before the beginning of the treatment, Time 2: after nine months from the beginning of active treatment.
  Lateral cephalometric images were taken for each patient, and this angle was measured in degrees.
Change in the UI- LI angle | Time 1: One week before the beginning of the treatment, Time 2: after nine months from the beginning of active treatment.
  Lateral cephalometric images were taken for each patient, and this angle was measured in degrees. This angle represents the relationship between the upper and the lower incisor axis in the cephalometric analysis in the anteroposterior direction.
Change in the NS-GN angle | Time 1: One week before the beginning of the treatment, Time 2: after nine months from the beginning of active treatment.
  Lateral cephalometric images were taken for each patient, and this angle was measured in degrees. This angle represents the growth pattern of the mandible in the cephalometric analysis in the vertical direction.
Change in the posterior facial height (S-Go) | Time 1: One week before the beginning of the treatment, Time 2: after nine months from the beginning of active treatment.
  Lateral cephalometric images were taken for each patient. This was measured in millimetres vertically from S point to GO point.
Change in the anterior facial height (N-Me) | Time 1: One week before the beginning of the treatment, Time 2: after nine months from the beginning of active treatment.
  Lateral cephalometric images were taken for each patient. This was measured in millimetres vertically from N point to Me point.
Change in the U1-Palatal plane measurement | Time 1: One week before the beginning of the treatment, Time 2: after nine months from the beginning of active treatment.
  Lateral cephalometric images were taken for each patient. This was measured in millimetres vertically from the upper central incisor apex and the palatal plane.
Change in the U6-Palatal plane measurement | Time 1: One week before the beginning of the treatment, Time 2: after nine months from the beginning of active treatment.
  Lateral cephalometric images were taken for each patient. This was measured in millimetres vertically from the tip of the mesial cusp of the upper first molar and the palatal plane.
Change in the L1-GoMe measurement | Time 1: One week before the beginning of the treatment, Time 2: after nine months from the beginning of active treatment.
  Lateral cephalometric images were taken for each patient. This was measured in millimetres vertically from the lower central incisor apex and the mandibular plane.
Change in the L6-GoMe measurement | Time 1: One week before the beginning of the treatment, Time 2: after nine months from the beginning of active treatment.
  Lateral cephalometric images were taken for each patient. This was measured in millimetres vertically from the tip of the mesial cusp of the lower first molar and the mandibular plane.

SECONDARY OUTCOMES:
Change in the Li-Esth measurement | Time 1: One week before the beginning of the treatment, Time 2: after nine months from the beginning of active treatment.
  Lateral cephalometric images were taken for each patient. This was measured in millimetres from the Labrale inferius and E-Line of Ricketts.
Change in the Ls-Esth measurement | Time 1: One week before the beginning of the treatment, Time 2: after nine months from the beginning of active treatment.
  Lateral cephalometric images were taken for each patient. This was measured in millimetres from the Labrale superius and E-Line of Ricketts.
Change in the Nasolabial angle | Time 1: One week before the beginning of the treatment, Time 2: after nine months from the beginning of active treatment.
  Lateral cephalometric images were taken for each patient, and this angle was measured in degrees. This angle represents the relationship between the nose and the upper lip in the cephalometric analysis in the anteroposterior direction.
Change in the Mentolabial angle | Time 1: One week before the beginning of the treatment, Time 2: after nine months from the beginning of active treatment.
  Lateral cephalometric images were taken for each patient, and this angle was measured in degrees. This angle represents the relationship between the chin and the lower lip in the cephalometric analysis in the anteroposterior direction.

CONTACTS AND LOCATIONS:
Overall Officials: Hammam Zeidan, DDS,MSc, Principal Investigator — Department of Orthodontics, University of Al-Baath Dental School, Hama, Syria.; Amjad A Hasan, DDS,MSc, Principal Investigator — Department of orthodontics, Damascus University, Syria; Mohammad Y. Hajeer, DDS,MSc,PhD, Study Director — Department of orthodontics, Damascus University, Syria; Azzam Al-Jundi, DDS,MSc,PhD, Study Director — Department of Orthodontics, University of Hama, Dental School, Hama, Syria.
Locations (1):
- University of Damascus, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pisani L, Bonaccorso L, Fastuca R, Spena R, Lombardo L, Caprioglio A. Systematic review for orthodontic and orthopedic treatments for anterior open bite in the mixed dentition. Prog Orthod. 2016 Dec;17(1):28. doi: 10.1186/s40510-016-0142-0. Epub 2016 Sep 19. PMID 27615261
- [Background] Feres MF, Abreu LG, Insabralde NM, de Almeida MR, Flores-Mir C. Effectiveness of open bite correction when managing deleterious oral habits in growing children and adolescents: a systematic review and meta-analysis. Eur J Orthod. 2017 Feb;39(1):31-42. doi: 10.1093/ejo/cjw005. Epub 2016 Feb 3. PMID 26846264
- [Background] Turkkahraman H, Cetin E. Comparison of two treatment strategies for the early treatment of an anterior skeletal open bite : Posterior bite block-vertical pull chin cup (PBB-VPC) vs. posterior bite block-high pull headgear (PBB-HPH). J Orofac Orthop. 2017 Jul;78(4):338-347. doi: 10.1007/s00056-017-0095-z. Epub 2017 May 9. PMID 28488080
- [Background] Meibodi SE, Fatahi Meybodi S, Samadi AH. The effect of posterior bite-plane on dentoskeletal changes in skeletal open-bite malocclusion. J Indian Soc Pedod Prev Dent. 2009 Oct-Dec;27(4):202-4. doi: 10.4103/0970-4388.57653. PMID 19915269
- [Background] Cinsar A, Alagha AR, Akyalcin S. Skeletal open bite correction with rapid molar intruder appliance in growing individuals. Angle Orthod. 2007 Jul;77(4):632-9. doi: 10.2319/071406-292. PMID 17605497